CLINICAL TRIAL: NCT05158764
Title: Evaluation of the Efficacy and Safety of the New URGO BD001 Compression System Versus a Reference Compression in the Local Treatment of Venous or Mixed Predominantly Venous Leg Ulcers: a Prospective Open-label RCT
Brief Title: Efficacy and Safety of URGOBD001 Compression System
Acronym: FUTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires URGO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID RCB : 2021-A01874-37
Record Dates: First submitted 2021-10-29; First posted 2021-12-15 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Venous Leg Ulcer
Keywords: compression system; VLU; mixed VLU
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- URGO BD001 (Experimental): Treatment with URGO DB001 during 12-week treament period (5 medical visits are planned: D0, W2, W4, W8, W12)
  Interventions: Device: Venous compression system of the lower limbs stage C6 / C6r of the CEAP classification
- Kit Biflex (Active Comparator): Treatment with Kit Biflex during 12-week treament period (5 medical visits are planned: D0, W2, W4, W8, W12
  Interventions: Device: Venous compression system of the lower limbs stage C6 / C6r of the CEAP classification

INTERVENTIONS:
Device: Venous compression system of the lower limbs stage C6 / C6r of the CEAP classification — Etiological treatment of venous disease of the lower limbs stage C6 / C6r
  Other Names: Etiological treatment of venous disease of the lower limbs stage C6 / C6r

SUMMARY:
Evaluation of the efficacy (wound epithelialization and time to closure) and safety (emergence and nature of adverse event) of the new URGO BD001 compression system versus a reference compression in the local treatment of venous or mixed predominantly venous leg ulcers: prospective multicenter, randomized controlled, open-label clinical study

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, open-label, multicenter clinical trial conducted in patients with a leg ulcer of venous or mixed predominantly venous origin of stage C6 / C6r of the CEAP classification.

This study is carried out in around 55 French investigational centers. A total of 178 patients meeting the eligibility criteria will be included. The patients will be followed for 12 weeks and a total of 5 clinical evaluations will be carried out by the investigating centers.

A planimetric survey of the studied VLU is carried out during the initial assessment of the wound (Day 0) and at each assessment provided for in the protocol (Week 2, Week 4, Week 8 and Week 12).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old), having given free, informed and written consent
* Patient affiliated to a social security scheme
* Patient agreeing to wear the study compression system daily
* Patient with an ankle circumference between 18 and 25 cm
* Target wound: stage C6 / C6r leg ulcer of the CEAP classification with a 0.8≤ ABPI≤1.3
* Target wound with an area between 1 and 20 cm2
* Target wound with age of ≤24 months

Criteria exclusion:

* Patient with a systemic infection not controlled by appropriate antibiotic therapy
* Patient having presented in the 3 months preceding his inclusion, a deep vein thrombosis
* Patient with advanced stage II or stage III lymphoedema
* Patient bedridden or spending less than an hour per day standing
* Clinically infected target wound
* Cancerized target wound

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Complete closure of the Venous Leg Ulcer (VLU) | 12-week treament period
  Complete closure of the leg ulcer is defined by 100% re-epithelialization of the Venous Leg Ulcer (VLU)

SECONDARY OUTCOMES:
Time to complete closure of the Venous Leg Ulcer (VLU) | 12-week treament period
  Time to complete closure of the Venous Leg Ulcer (VLU) is defined as the time from inclusion to the date of complete closure
Safety analysis | 12-week treament period
  Nature and number of adverse event related to the use of the studied compression system (serious/ non-serious)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Dr SENET, MD, Principal Investigator — Hôpitaux Universitaires Paris Est (AP-HP) - Hopital TENON
Locations (1):
- Patricia SENET, Paris, France

IPD SHARING:
Plan to Share IPD: No